CLINICAL TRIAL: NCT01975272
Title: The Value of Iron Treatment for Postoperative Obstetric Patients With Anemia: a Randomized Double Blind Controlled Trial
Brief Title: The Use of Iron Therapy for Patients With Anemia After Caesarean Section
Acronym: VITAPOP
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Disapointing randomization rate
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Vifor Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: METC 12-2-018
Record Dates: First submitted 2013-09-30; First posted 2013-11-04 (Estimated); Results first posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-03

CONDITIONS: Postoperative Anaemia
Keywords: postoperative; anemia; gynaecologic; surgery
MeSH Terms: conditions — Anemia | interventions — ferric carboxymaltose; ferrous fumarate; Iron; Fumarates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ferinject (Active Comparator): Once an infusion of Ferinject 1000 mg, 1 day after surgery
  Interventions: Drug: Ferinject; Drug: Placebo for ferrous fumarate
- Ferrous fumarate (Active Comparator): 2 times a day 200 mg ferrous fumarate, starting 24-48 hours after surgery
  Interventions: Drug: Ferrous fumarate; Drug: Placebo for ferinject
- Placebo infusion and tablets (Placebo Comparator): Patient will get a once a placebo infusion (250 ml NaCl), one day after surgery, and 60 placebo tablets for 30 days (2 tablets a day), starting 24-48 hours after surgery
  Interventions: Drug: Placebo for ferrous fumarate; Drug: Placebo for ferinject

INTERVENTIONS:
Drug: Ferinject
  Other Names: intravenous iron; ferric carboxymaltose
  Arms: Ferinject
Drug: Ferrous fumarate
  Other Names: Oral iron; Iron (II) fumarate
  Arms: Ferrous fumarate
Drug: Placebo for ferrous fumarate
  Other Names: Placebo tablets
  Arms: Ferinject; Placebo infusion and tablets
Drug: Placebo for ferinject
  Other Names: NaCl
  Arms: Ferrous fumarate; Placebo infusion and tablets

SUMMARY:
The purpose of this study is to determine whether oral or intravenous iron is effective in the treatment of anaemia (iron-poor blood) after caesarean section.

DETAILED DESCRIPTION:
Anemia after caesarean section is often treated with iron therapy to ensure that the hemoglobin will return to normal more rapidly. Scientific evidence for this action is limited. Several studies, in which iron therapy was given after orthopaedic or cardiac surgery, show that after 6 to 10 weeks the hemoglobin was not significantly different between patients treated with oral preparations and patients treated with a placebo. These studies have not examined the hemoglobin level during the first few weeks after surgery including the quality of life analysis.

The purpose of this double blind randomized controlled trial therefore is to examine the effect of both oral iron therapy and intravenous iron therapy on hemoglobin level and on the quality of life during the first few weeks postcaesarean in patients with a moderate anemia.

ELIGIBILITY:
Inclusion Criteria:

* Gynecological surgery
* Hb 5-7 mmol/L

Exclusion Criteria:

* Pregnancy
* Oncological operations
* Infections (PID)
* Diagnostic procedures: level 1 laparoscopies (diagnostic, sterilization, tubal testing; Hysteroscopies
* Smaller therapeutic procedures: large loop excision of transformation zone (LLETZ), Conization,
* Small vulvar / vaginal operations such as (cysts, labia correction)
* Endometrial ablation
* Legal incapacity
* The patient has used pre-operatively an iron preparation and / or blood transfusion or during the surgery
* Hematologic disorders
* Erythropoiesis-stimulating agents < 3months ago
* Myelosuppressive therapy in history
* Hepatitis
* HIV
* Alcohol abuses
* Not understanding Dutch
* Allergic reaction to iron therapy in past

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-03-02 (Actual); Primary Completion 2018-05-17 (Actual); Study Completion 2018-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy Kruitwagen, Principal Investigator — Maastricht University Medical Center
Locations (2):
- Netherlands (2):
  - Maastricht University Medical Centre, Maastricht, Limburg
  - Orbis Medical Centre, Sittard, Limburg

RESULTS

PARTICIPANT FLOW:
Groups:
- Ferinject: Once an infusion of Ferinject 1000 mg, 1 day after surgery
  Ferinject
  Placebo for ferrous fumarate
- Ferrous Fumarate: 2 times a day 200 mg ferrous fumarate, starting 24-48 hours after surgery
  Ferrous fumarate
  Placebo for ferinject
- Placebo Infusion and Tablets: Patient will get a once a placebo infusion (250 ml NaCl), one day after surgery, and 60 placebo tablets for 30 days (2 tablets a day), starting 24-48 hours after surgery
  Placebo for ferrous fumarate
  Placebo for ferinject
Period: Overall Study
Arm/Group | Ferinject | Ferrous Fumarate | Placebo Infusion and Tablets
Started | 9 | 10 | 8
Completed | 8 | 9 | 6
Not Completed | 1 | 1 | 2
Not completed — Excluded after protocol amendment | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: A significant number of patients were lost to follow-up: 2 patients Ferinject group, 4 patients Ferrous fumarate group, and 2 patients placebo group.
  Most likely reason: no complaints in a phase in which attention to the newborn was given priority.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ferinject | Ferrous Fumarate | Placebo Infusion and Tablets | Total
Number analyzed (Participants) | 8 | 9 | 6 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 6 | 23
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 6 | 23
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 8 | 9 | 6 | 23

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin
Description: Serum hemoglobin level
Time Frame: 3 weeks postoperative
Measure: Mean (Full Range); unit: mmol/L
Arm/Group | Ferinject | Ferrous Fumarate | Placebo Infusion and Tablets
Number analyzed (Participants) | 6 | 5 | 4
mmol/L | 8.4 [7.8 to 8.8] | 7.9 [7.4 to 8.0] | 7.1 [7.1 to 7.4]

2. Secondary Outcome: Serum Ferritin
Description: Serum levels of ferritin
Time Frame: 3 weeks postoperative
Measure: Mean (Full Range); unit: microgram/L
Arm/Group | Ferinject | Ferrous Fumarate | Placebo Infusion and Tablets
Number analyzed (Participants) | 6 | 5 | 4
microgram/L | 422 [21 to 682] | 57 [29 to 125] | 37 [14 to 80]

3. Secondary Outcome: Serum Hepcidin
Description: Serum hepcidin level
Time Frame: 3 weeks postoperative
Measure: Mean (Full Range); unit: nmol/L
Arm/Group | Ferinject | Ferrous Fumarate | Placebo Infusion and Tablets
Number analyzed (Participants) | 6 | 5 | 4
nmol/L | 11.6 [0.5 to 25.7] | 2.2 [0.5 to 5.2] | 1.7 [0.5 to 4.6]

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Ferinject | Ferrous Fumarate | Placebo Infusion and Tablets
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 0/9 | 0/10 | 0/8

LIMITATIONS AND CAVEATS:
Evident conclusions cannot be drawn from this small prematurely stopped study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-09): https://cdn.clinicaltrials.gov/large-docs/72/NCT01975272/Prot_SAP_000.pdf